CLINICAL TRIAL: NCT06696079
Title: Restarting Early Versus Later Anticoagulation for Chronic Subdural Hematoma With Atrial Fibrillation (RELACS): An International Multicenter, Randomized Controlled, Two-arm, Assessor-blinded, Trial
Brief Title: Restarting Early Versus Later Anticoagulation for Chronic Subdural Hematoma With Atrial Fibrillation
Acronym: RELACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rahul Raj (Other)
Collaborators: Tampere University Hospital (Other); Kuopio University Hospital (Other); Turku University Hospital (Other Government); Oulu University Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Sponsor-Investigator, Rahul Raj, Sponsor Principal Investigator, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUS/7351/2024
Record Dates: First submitted 2024-11-18; First posted 2024-11-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2024-11

CONDITIONS: Chronic Subdural Hematoma; Atrial Fibrillation (AF)
Keywords: chronic subdural hematoma; atrial fibrillation; oral anticoagulation; warfarin; direct oral anticoagulants; surgery; stroke; hemorrhage; prognosis
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Atrial Fibrillation; Stroke; Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor masking and blinded data interpretation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early resumption (Experimental): Oral anticoagulation therapy is resumed on the 5th postoperative day following burr-hole surgery for chronic subdural hematoma.
  Interventions: Drug: Early Resumption of Oral Anticoagulation Therapy
- Late resumption (Active Comparator): Oral anticoagulation therapy is resumed on the 30th postoperative day following burr-hole surgery for chronic subdural hematoma.
  Interventions: Drug: Late Resumption of Oral Anticoagulation Therapy

INTERVENTIONS:
Drug: Early Resumption of Oral Anticoagulation Therapy — The patient's prescribed anticoagulant therapy for atrial fibrillation is resumed on the 5th postoperative day following burr-hole surgery for chronic subdural hematoma. This early resumption strategy is compared to the standard practice of resuming anticoagulation therapy on the 30th postoperative day.
  Arms: Early resumption
Drug: Late Resumption of Oral Anticoagulation Therapy — The patient's prescribed anticoagulant therapy for atrial fibrillation is resumed on the 30th postoperative day following burr-hole surgery for chronic subdural hematoma. This standard resumption strategy is compared to the early approach of resuming anticoagulation therapy on the 5th postoperative day.
  Arms: Late resumption

SUMMARY:
The goal of this randomized clinical trial is to assess the benefit of early resumption versus late resumption of oral anticoagulation medication in adults with atrial fibrillation undergoing surgery for chronic subdural hematoma. The main questions it aims to answer are:

* Does anticoagulation resumption 5 days after surgery as compared to 30 days after surgery result in fewer thromboembolic complications, without increasing the risk for bleeding?
* Does anticoagulation resumption 5 days after surgery as compared to 30 days after surgery affect the risk of reoperation, functional outcome, mortality, and healthcare use?

Researchers will compare early anticoagulation resumption (5 days) and late anticoagulation resumption (30 days) after chronic subdural hematoma surgery.

Participants will either resume the medication 5 days or 30 days after the surgery. The participants will be followed up for 3 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Patients with a symptomatic unilateral or bilateral CSDH requiring burr-hole evacuation with drainage (CSDH is predominantly hypodense or isodense on imaging [CT/MRI]; clinical symptoms attributable to the CSDH; patients with bilaterally operated CSDHs will be treated with the same protocol on both sides and analyzed as a single study participant).
* Patients that are on an oral anticoagulation medication due to permanent, persistent or paroxysmal spontaneous atrial fibrillation previously known
* Randomization done within 4 days of the surgery

Exclusion Criteria:

* Intraoperative or immediate postoperative hemorrhagic complication
* CSDH requiring surgical treatment other than burr-hole evacuation (e.g. craniotomy)
* Prior CSDH surgery within 12 months
* Cerebrospinal fluid shunt
* CSDH is in an arachnoid cyst
* If the operated hematoma is revealed to be a cerebrospinal fluid collection (hygroma)
* Conditions other than atrial fibrillation that require anticoagulation, including therapeutical dose of low molecular-weight heparin or heparin (for example, pulmonary embolism, deep vein thrombosis, hypercoagulability syndromes)
* Mechanical heart valve(s)
* Moderate or severe mitral stenosis (other valvular diseases and biological valves are eligible)
* Contraindication to anticoagulation medication (for example bleeding disorder, documented high risk of fall [e.g. due to severe alcoholism], severe thrombocytopenia, severe anemia)
* Concomitant use of antiplatelet medication
* Moderate to severe renal insufficiency (creatinine clearance <30 ml/min or on dialysis)
* Not a permanent resident in Finland (for Finnish patients) or not a permanent resident in Region Stockholm (for Swedish patients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 332 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Rate of composite outcome of vascular events | 90 days
  Rate of the composite outcome that combines thromboembolic events (ischemic stroke, systemic embolism), hemorrhagic events (intracranial hemorrhage, major extracranial bleeding), and vascular death.

SECONDARY OUTCOMES:
Rate of different components of the primary composite outcome | 90 days
  Separation of the components of the primary composite outcome (thromboembolic, hemorrhagic, vascular death).
Rate of patients with favorable functional outcome | 90 days
  Assessed using the modified Rankin Scale (mRS), which ranges from 0 (no symptoms) to 6 (death).
Rate of reoperation | 90 days
  Reoperation for the initially treated chronic subdural hematoma.
Rate of all-cause mortality | 90 days and 12 months
Participants' healthcare use | 90 days
  Number and type of unscheduled emergency radiological examinations, - number of emergency department visits, postoperative total hospitalization days

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Raj, MD, PhD, Study Chair — Helsinki University Hospital & University of Helsinki; Jarno Satopää, MD, PhD, Principal Investigator — Helsinki University Hospital & University of Helsinki; Jussi P Posti, MD, PhD, Principal Investigator — Turku University Hospital and University of Turku; Teemu Luoto, MD, PhD, Principal Investigator — Tampere University Hospital and Tampere University; Nils Danner, MD, PhD, Principal Investigator — Kuopio University Hospital and University of Eastern Finland; Oula Knuutinen, MD, PhD, Principal Investigator — Oulu University Hospital and University of Oulu; Jiri Bartek, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (6):
- Finland (5):
  - Oulu University Hospital, Oulu, North Ostrobothnia
  - Kuopio University Hospital, Kuopio, Northern Savonia
  - Tampere University Hospital, Tampere, Pirkanmaa
  - Turku University Hospital, Turku, Southwest Finland
  - Helsinki University Hospital, Helsinki, Uusimaa
- Karolinska University Hospital, Stockholm, Region Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Researcher-initiated data sharing is not possible due to the Finnish Secondary Use Act (552/2019). Thus, all requests to process data for purposes permitted by the Secondary Use Act are given based on an official decision made by FINDATA (https://findata.fi/en/).